CLINICAL TRIAL: NCT02258477
Title: A Pilot Study: Snacking, Willpower and Glucose Availability
Acronym: SWG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 14-1485
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Willpower
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (D-B-A-C) (Active Comparator): 100 calorie beverage during week 1; 10 calorie beverage during week 2; control beverage beverage during week 3; 50 calorie beverage during week 4.
  Interventions: Dietary Supplement: Sequence 1
- Sequence 2 (A-D-C-B) (Active Comparator): Control beverage during week 1; 100 calorie beverage during week 2; 50 calorie beverage during week 3; 10 calorie beverage during week 4.
  Interventions: Dietary Supplement: Sequence 2
- Sequence 3 (C-A-B-D) (Active Comparator): 50 calorie beverage during week 1; control beverage during week 2; 10 calorie beverage during week 3; 100 calorie beverage during week 4.
  Interventions: Dietary Supplement: Sequence 3
- Sequence 4 (B-C-D-A) (Active Comparator): 10 calorie beverage during week 1; 50 calorie beverage during week 2; 100 calorie beverage during week 3; control beverage during week 4.
  Interventions: Dietary Supplement: Sequence 4

INTERVENTIONS:
Dietary Supplement: Sequence 1 — 100 calorie beverage during week 1; 10 calorie beverage during week 2; control beverage beverage during week 3; 50 calorie beverage during week 4.
  Arms: Sequence 1 (D-B-A-C)
Dietary Supplement: Sequence 2 — Control beverage during week 1; 100 calorie beverage during week 2; 50 calorie beverage during week 3; 10 calorie beverage during week 4.
  Arms: Sequence 2 (A-D-C-B)
Dietary Supplement: Sequence 3 — 50 calorie beverage during week 1; control beverage during week 2; 10 calorie beverage during week 3; 100 calorie beverage during week 4.
  Arms: Sequence 3 (C-A-B-D)
Dietary Supplement: Sequence 4 — 10 calorie beverage during week 1; 50 calorie beverage during week 2; 100 calorie beverage during week 3; control beverage during week 4.
  Arms: Sequence 4 (B-C-D-A)

SUMMARY:
To compare the effects of ingesting 100, 50 and 10 calories of glucose as compared to a non-calorie placebo (0 calorie beverage) on self-control over resisting snack foods. To test whether there is a threshold of glucose that will result in improved ease of resistance to problem foods (tested by comparing three different levels of glucose).

DETAILED DESCRIPTION:
Ingestion of 100 calories of glucose during individually pre-determined times of waning dietary self-control will result in improved ease of resistance to problem foods when compared to ingestion of lower calories of glucose or placebo (0 calorie beverage)

ELIGIBILITY:
Inclusion Criteria:

1. Females ages 18 - 65 years.
2. Self-identify as regular snackers, with a specific problem food, who have trouble with over-consuming this snack food.
3. Have intentionally lost weight in the last year and are seeking to maintain that weight loss or have unintentionally gained weight in the last year and are concerned about it.
4. Generally healthy.

Exclusion Criteria:

1. Pregnant or trying to become pregnant.
2. Diagnosis of type 1 or type 2 diabetes
3. Not willing or able to follow study guidelines (ie: consuming the study beverage daily for four weeks, or completing daily compliance logs)
4. Current smoker (or has stopped smoking within the last 6 months)
5. Taking medications that could cause weight loss or weight gain (such as steroids, tricyclic antidepressants, chemotherapy, antipsychotics, prescribed or over the counter weight loss agents, etc).
6. Current or history of eating disorder (anorexia, bulimia, or diagnosed binge eating disorder)
7. Current alcohol or drug abuse or dependence
8. Any medical condition for which daily snacking of such problem foods would be inadvisable (i.e.: a subject with hypertension advised to avoid sodium).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James O Hill, PhD, Principal Investigator — Anschutz Health and Wellness Center
Locations (1):
- Anschutz Health and Wellness Center, Aurora, Colorado, United States

REFERENCES:
- [Background] Hand GA, Shook RP, Paluch AE, Baruth M, Crowley EP, Jaggers JR, Prasad VK, Hurley TG, Hebert JR, O'Connor DP, Archer E, Burgess S, Blair SN. The energy balance study: the design and baseline results for a longitudinal study of energy balance. Res Q Exerc Sport. 2013 Sep;84(3):275-86. doi: 10.1080/02701367.2013.816224. PMID 24261006
- [Background] Chang SH, Pollack LM, Colditz GA. Life Years Lost Associated with Obesity-Related Diseases for U.S. Non-Smoking Adults. PLoS One. 2013 Jun 18;8(6):e66550. doi: 10.1371/journal.pone.0066550. Print 2013. PMID 23823705
- [Background] Dulloo AG. Explaining the failures of obesity therapy: willpower attenuation, target miscalculation or metabolic compensation? Int J Obes (Lond). 2012 Nov;36(11):1418-20. doi: 10.1038/ijo.2012.114. No abstract available. PMID 23147189
- [Background] Masicampo EJ, Baumeister RF. Toward a physiology of dual-process reasoning and judgment: lemonade, willpower, and expensive rule-based analysis. Psychol Sci. 2008 Mar;19(3):255-60. doi: 10.1111/j.1467-9280.2008.02077.x. PMID 18315798
- [Background] Littell, Ramon C., George A. Milliken, Walter W. Stroup, Russell D. Wolfinger, and O Schabenberger. 2006. SAS@ for Mixed Models, Second Edition. Cary, NC: SAS Institute.
- [Result] Gailliot MT, Baumeister RF. The physiology of willpower: linking blood glucose to self-control. Pers Soc Psychol Rev. 2007 Nov;11(4):303-27. doi: 10.1177/1088868307303030. PMID 18453466
- [Result] Hofmann W, Adriaanse M, Vohs KD, Baumeister RF. Dieting and the self-control of eating in everyday environments: an experience sampling study. Br J Health Psychol. 2014 Sep;19(3):523-39. doi: 10.1111/bjhp.12053. Epub 2013 Jun 10. PMID 23751109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using study flyers and the study was posted on the Center website.
Pre-assignment Details: Note, that each subject participated in the study for four weeks, consuming a different study beverage daily for one week, being crossed-over to another beverage the following week. Thus a total of 33 subjects completed all four weeks of the cross-over study.
Groups:
- Sequence 1 (D-B-A-C): Subjects assigned to sequence 1 received 100 calorie beverage in week 1, 10 calorie beverage in week 2, 0 calorie control beverage in week 3, and 50 calorie beverage in week 4.
- Sequence 2 (A-D-C-B): Subjects in sequence 2 received 0 calorie control beverage in week 1, 100 calorie beverage in week 2, 50 calorie beverage in week 3, and 10 calorie beverage in week 4.
- Sequence 3 (C-A-B-D): Subjects in sequence 3 received 50 calorie beverage in week 1, 0 calorie control beverage in week 2, 20 calorie beverage in week 3, and 100 calorie beverage in week 4.
- Sequence 4 (B-C-D-A): Subjects in sequence 4 received 10 calorie beverage in week 1, 50 calorie beverage in week 2, 100 calorie beverage in week 3, and 0 calorie control beverage in week 4.
Period: First Intervention (1 Week)
Arm/Group | Sequence 1 (D-B-A-C) | Sequence 2 (A-D-C-B) | Sequence 3 (C-A-B-D) | Sequence 4 (B-C-D-A)
Started | 10 | 9 | 9 | 9
Completed | 9 | 8 | 9 | 9
Not Completed | 1 | 1 | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Sequence 1 (D-B-A-C) | Sequence 2 (A-D-C-B) | Sequence 3 (C-A-B-D) | Sequence 4 (B-C-D-A)
Started | 9 | 8 | 9 | 9
Completed | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 1 | 1
Period: Third Intervention (1 Week)
Arm/Group | Sequence 1 (D-B-A-C) | Sequence 2 (A-D-C-B) | Sequence 3 (C-A-B-D) | Sequence 4 (B-C-D-A)
Started | 9 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention (1 Week)
Arm/Group | Sequence 1 (D-B-A-C) | Sequence 2 (A-D-C-B) | Sequence 3 (C-A-B-D) | Sequence 4 (B-C-D-A)
Started | 9 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 37 subjects were screened and enrolled into the study. Each subject was randomized to a different sequence of consumption of the weekly study beverage. 33 subjects completed the 4 week study.
Groups:
- All Study Subjects: Compare the efficacy of 0 calorie sucralose-sweetened water on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Glucose: This is a randomized, double-blind cross-over pilot study involving 40 study subjects. We will compare the efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food. After baseline data collection, eligible participants will be randomized into one of the four sequence group and receive a different beverage each week.
Arm/Group | All Study Subjects
Number analyzed (Participants) | 37
Age, Customized [Mean (Standard Deviation); unit: years] | 44.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 24
  More than one race | 3
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Responses to the Control of Eating Questionnaire
Description: Study participant will complete Eating Questionnaire at baseline and the next 4 visits. Each questionnaire item used a likert scale (with ratings from 1 - 10). All question pertain to the last 7 days. Questionnaire items #9 asked "what one food makes it most difficult for you to control eating?" and question #10 asked " What time are you particularly vulnerable to this one food." Higher ratings are consistent with a more significant or more frequent outcome.
  Note that values in the data table below are absolute scores at each week that the subject consumed the noted treatment dose. As subjects were randomized to different sequence orders to receive the study beverages, subjects consumed any given treatment dose at different weeks (depending on their randomized sequence order).
Time Frame: 4 weeks
Population: 33 participants completed the 4 week study and were randomized to one of four treatment sequences. Thus, each subject received each treatment for one week.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Compare the efficacy of 0 calorie sucralose-sweetened water on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence groups and received each treatment for 1 week.
- 100 Calorie Glucose Beverage: Compare the efficacy of a 100 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence group and receive each treatment for 1 week.
- 50 Calorie Beverage: Compare the efficacy of a 50 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence groups and received each treatment for 1 week.
- 10 Calorie: Compare the efficacy of a 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence groups and received each treatment for 1 week.
Arm/Group | Control | 100 Calorie Glucose Beverage | 50 Calorie Beverage | 10 Calorie
Number analyzed (Participants) | 33 | 33 | 33 | 33
units on a scale
  Question 1: frequency of food cravings | 4.5 (2.1) | 5.2 (2.7) | 5.1 (2.4) | 5.2 (2.4)
  Question 2: strength of cravings | 4.6 (2.3) | 5.0 (2.6) | 4.8 (2.6) | 5.1 (2.4)
  Question 3: difficulty to resisit cravings | 4.3 (2.5) | 5.2 (2.8) | 5.0 (2.6) | 5.5 (2.7)
  Question 4: frequency of eating due to cravings | 4.2 (1.8) | 4.8 (2.6) | 5.1 (2.4) | 4.9 (2.1)
  Question 5: Freq of cravings for chocolate | 3.6 (2.4) | 4.0 (2.7) | 3.9 (2.6) | 4.6 (2.6)
  Question 6: Freq of cravings for other sweet foods | 3.8 (2.6) | 4.5 (2.8) | 4.5 (2.8) | 4.6 (2.8)
  Question 7: Freq of cravings for fruit | 2.5 (1.7) | 2.9 (2.0) | 2.7 (1.8) | 2.9 (1.6)
  Question 8: Freq of cravings for savory foods | 4.1 (2.1) | 4.3 (2.3) | 4.6 (2.3) | 4.7 (2.4)
  Question 11: Freq of eating problem food | 4.9 (2.6) | 4.9 (3.2) | 4.6 (2.9) | 4.8 (2.8)
  Question 12: Difficulty resisting problem food | 5.1 (2.5) | 6.4 (3.1) | 5.5 (2.9) | 6.2 (2.7)
  Question 13: Difficulty controlling eating | 4.6 (1.8) | 5.8 (2.9) | 5.9 (2.5) | 5.5 (2.2)
  Question 14: Freq of snacking | 5.5 (2.4) | 6.0 (2.8) | 6.1 (2.5) | 6.3 (2.3)
  Question 15: Freq of skipping meals | 3.0 (1.9) | 2.8 (2.0) | 2.8 (1.7) | 2.9 (1.8)
  Question 16: Frequency of eating alone | 5.3 (2.8) | 5.0 (2.8) | 5.4 (2.7) | 5.4 (2.5)
  Question #17: Freq of eating alone | 5.9 (2.5) | 6.2 (2.8) | 5.7 (2.5) | 5.9 (2.7)
  Question 18: Freq of eating while doing other | 5.9 (2.4) | 5.8 (2.6) | 5.6 (2.2) | 6.0 (2.4)
  Question 19: Freq of eating more than intended | 3.9 (2.2) | 4.7 (2.5) | 4.7 (2.6) | 4.7 (2.3)
  Question 20: Freq of watching calories/portions | 5.7 (2.6) | 5.6 (3.2) | 5.4 (2.7) | 5.6 (2.9)

2. Secondary Outcome: Number of Days That a Problem Snack Food Was Consumed at the Identified Time of Waning Dietary Self-control.
Description: Study participant will record if the problem snack was consumed each day within the 3 hour period following consumption of the study beverage.
  Note that the values in the data table below reflect the percentage of days within a week that subjects within each treatment dose consumed a problem snack food at the identified time of waning dietary self-control. The data does not represent change from baseline, but rather percentage of days within a week (calculated by how many days within a week subject consumed the problem snack food at the identified time of waning dietary self-control/ 7 days in a week) and can be compared week by week to see if there is any significant difference weekly when consuming a different dose of glucose.
Time Frame: 4 weeks
Population: 33 subjects completed the 4 week study.
Measure: Mean (Standard Deviation); unit: percentage of days in a week
Groups:
- 50 cal Glucose Beverage: Compare the efficacy of a 50 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence groups and received each treatment for 1 week.
- 10 cal Glucose Beverage: Compare the efficacy of a 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food.
  Efficacy of a 100, 50, and 10 calorie glucose beverage versus an identical volume of placebo beverage (0 calorie sucralose-sweetened water) on the behavioral ease of resisting problem foods during time of vulnerability to the problem food was compared. After baseline data collection, eligible participants were randomized into one of the four sequence groups and received each treatment for 1 week.
Arm/Group | Control | 100 Calorie Glucose Beverage | 50 cal Glucose Beverage | 10 cal Glucose Beverage
Number analyzed (Participants) | 33 | 33 | 33 | 33
percentage of days in a week | 13.3 (14.2) | 16.0 (18.8) | 14.6 (20.0) | 14.1 (16.7)

3. Secondary Outcome: Number of Days That a Problem Snack Food Was Consumed at Any Time of Day in a Week.
Description: Study participant will record daily the time problem snack food was consumed. Note that the values in the data table below reflect the percentage of days within a week that subjects within each treatment dose consumed a problem snack food at any time of day. The data does not represent change from baseline, but rather percentage of days within a week (calculated by how many days within a week subject consumed the problem snack food at any time of day/ 7 days in a week) and can be compared week by week to see if there is any significant difference weekly when consuming a different dose of glucose.
Time Frame: 4 weeks
Population: 33 subjects completed the 4 week study.
Measure: Mean (Standard Deviation); unit: percentage of days in a week
Arm/Group | Control | 100 Calorie Glucose Beverage | 50 cal Glucose Beverage | 10 cal Glucose Beverage
Number analyzed (Participants) | 33 | 33 | 33 | 33
percentage of days in a week | 41.3 (23.6) | 44.1 (30.5) | 41.0 (28.0) | 43.3 (27.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the four-week study for each study participant.
Description: Adverse events were collected without regard for the intervention that was being administered.
Groups:
- All Study Subjects: Subjects were randomized into four possible sequences: subjects assigned to sequence 1 received the control beverage first during week 1, then the 10 calorie beverage during week 2, then the 50 calorie beverage during week 3, and then the 100 calorie beverage during week 4. Subjects assigned to sequence 2 received received the 50 calorie beverage during week 1, then the 100 calorie beverage during week 2, then the control beverage during week 3, and then the 50 calorie beverage during week 4. Subejcts assigned to sequence 3 received the 50 calorie beverage during week 1, then the control beverage during week 2, then the 100 calorie beverage during week 3, and then the 10 calorie beverage during week 4. Subjects assigned to sequence 4 received the 100 calorie beverage during week 1, then the 50 calorie beverage during week 2, then the 10 calorie beverage during week 3, and then the control beverage during week 4.
Arm/Group | All Study Subjects
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 9/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Subjects (N=37)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
fever (General disorders) | 1 (1)
migraine (General disorders) | 1 (1)
stomach ache (Gastrointestinal disorders) | 1 (1)
jitteriness (General disorders) | 1 (1)
Flu (General disorders) | 1 (1)
bursitis (Musculoskeletal and connective tissue disorders) | 1
dry mouth (General disorders) | 1 (1)
upset stomach (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
bloating (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study questionnaire involved limitations as questions were subjective in terms of how subjects defined cravings and snacking behavior. Also, food diaries may not be fully accurate accounts of subjects' actual caloric intake and food consumption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No